CLINICAL TRIAL: NCT04478903
Title: Perceived Burden and Quality of Life of Primary Caregivers of Cancer Patients Aged 70 and Older After 5 Years of Management
Acronym: FARAPPAC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: QUIPOURT 2019
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Quality of Life; Primary Patient Caregiver; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- primary caregiver of patients aged 70 and over
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Zarit Burden Inventory French version and SF12

SUMMARY:
Cancer is a disease that requires long-term management, especially now that medical advances have transformed most cancers from an acute to a chronic condition. Most of the time, therefore, the help provided by family and friends is long-term.

The negative impact of oncological care on the quality of life of family caregivers has already been studied. The UCOGB carried out a study in 2014 on the primary caregivers of cancer patients aged 70 and over at inclusion and at 3 and 6 months of oncogeriatric care. This study showed that several factors were significantly related to the caregiver's quality of life: the caregiver's age, perception of burden and patient autonomy (18). However, the evolution of quality of life and burden at 5 years has, to our knowledge, never been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Person who does not object to being included in the study
* Primary caregiver of a cancer patient aged 70 years and over who is managed in one of the centres participating in the study, with a request for an oncogeriatric consultation between 01/06/2014 and 18/03/2015.
* Age ≥ 18 years old
* Good command of the French language

Exclusion Criteria:

* Refusal or linguistic or psychological inability to answer the questionnaires.
* Caregiver whose general condition does not allow him/her to answer a questionnaire
* Death of the caregiver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrieval of information and contact details of primary caregivers included in the 2014 study along with the patient's vital status
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
To determine the quality of life of the primary caregiver of cancer patients 70 years of age and older, 5 years after initial management. | Through study completion, an average of 1 year
  Quality of life is measured using the SF-12 (short form) questionnaire. This is an abbreviated version of the Medical Outcomes Study Short-form General Health survey (SF-36).

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Derived] Barben J, Billa O, Collot J, Collot T, Manckoundia P, Bengrine-Lefevre L, Dabakuyo-Yonli TS, Quipourt V. Quality of life and perceived burden of the primary caregiver of patients aged 70 and over with cancer 5 years after initial treatment. Support Care Cancer. 2023 Feb 2;31(2):147. doi: 10.1007/s00520-023-07594-w. PMID 36729239